CLINICAL TRIAL: NCT06969768
Title: Integrative Multi-Omics Refines the Molecular Subtypes of Thyroid Cancers and Enhances Cancer-Progression Prediction
Brief Title: Proteogenomics for Follicular Cell-derived Thyroid Cancer: Development of a Classification and Prognosis Prediction Model
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government); National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, YoungJoo Park, Professor, Seoul National University Hospital
Other Study IDs: 1802-067-922
Record Dates: First submitted 2025-04-30; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Thyroid Cancer
Keywords: Thyroid cancer; Proteogenomics
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Surgical specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thyroid cancer: All patients diagnosed with thyroid cancer who underwent thyroidectomy at Seoul National University Hospital

SUMMARY:
This study aims to refine the molecular classification of thyroid cancer (TC) using a multi-omics approach. By identifying a novel gene set and applying decision-tree modeling, the study seeks to improve diagnostic accuracy and predict tumor progression in BRAFV600E-like and RAS-like TC subtypes. Protein biomarkers were validated via immunohistochemistry (IHC), with findings confirmed across external datasets.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed clinical diagnosis of thyroid cancer
* Availability of surgically resected thyroid tissue suitable for omics analysis

Exclusion Criteria:

- Patients who have received chemotherapy for other malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with thyroid cancer
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Classification Accuracy of Gene-Based Model | 1 year
  The accuracy of the decision-tree model using specific gene set to classify thyroid cancer into BRAFV600E-like, RAS-like, and NT (normal thyroid) -like subtypes. Model performance will be evaluated using accuracy, sensitivity, specificity, and Cohen's kappa.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea